CLINICAL TRIAL: NCT03355001
Title: Assessment of the Performance of Monosyn® Quick Suture Material in Different Indications Under Daily Clinical Routine.
Brief Title: Prospective, International Monosyn® Quick - Non Interventional Study
Acronym: PRIMOQ
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1635
Record Dates: First submitted 2017-10-26; First posted 2017-11-28 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Pediatric and Adult: Mucosal Closure in Facial and Oral Surgery; Pediatric and Adult: Skin Closure (Dermal Sutures); Women: Episiotomy; Pediatric: Urological Interventions (Circumcision, Phimosis Etc.)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Skin Closure: Monosyn® Quick will be used for skin closure for the adaptation of soft tissue and mucous membranes, when wound support over a period of 7 days is considered adequate.
  Interventions: Device: Monosyn® Quick
- Urology: Monosyn® Quick will be used in urology for the adaptation of soft tissue and mucous membranes, when wound support over a period of 7 days is considered adequate.
  Interventions: Device: Monosyn® Quick
- Gynecology: Monosyn® Quick will be used in gynecology for the adaptation of soft tissue and mucous membranes, when wound support over a period of 7 days is considered adequate.
  Interventions: Device: Monosyn® Quick

INTERVENTIONS:
Device: Monosyn® Quick — * Mucosal sutures in the facial and oral
  * Dermal sutures, particularly in pediatrics
  * Episiotomy
  * Circumcision

SUMMARY:
The Monosyn® Quick non-interventional study (NIS) has been designed to implement an action within the framework of a proactive post-market surveillance system.

The aim of this NIS is to collect systematically and proactively different clinical parameters regarding safety, effectiveness and performance of Monosyn® Quick suture material under the daily clinical practice when used as intended.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and adult patients undergoing mucosal wound or skin closure using Monosyn® Quick as suture material or women undergoing an episiotomy or pediatric patients undergoing an urological intervention such as a circumcision or phimosis or hypospadias etc.
* Written informed regarding the data collection for the Post Market Clinical Follow-Up (PMCF)

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult patients undergoing mucosal wound or skin closure using Monosyn® Quick as suture material or women undergoing an episiotomy or pediatric patients undergoing an urological intervention as a circumcision or phimosis or hypospadias
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-21 (Actual)

PRIMARY OUTCOMES:
Complication | at follow-up visit depending on routine clinical practice (approx. 1-3 months postoperatively)
  Descriptive Analysis of the Frequency of tissue reaction or inflammation, wound infection, seroma, fistula, abscess formation, hematoma, suture removal or re-suturing at different time points

SECONDARY OUTCOMES:
Complications | until day of discharge (approximately 1 week)
  Descriptive Analysis of dehiscence rates of the skin needing surgical treatment with re-closure
Dehiscence | until day of discharge (approximately 1 week) and at follow-up visit depending on routine clinical practice (approx. 1-3 months postoperatively)
  Descriptive Analysis of dehiscence rates of the skin needing surgical treatment with re-closure for two different intervals: time of Intervention until day of discharge as well as day of discharge until follow-up visit at approximately 1-3 months postoperatively
Patient and Observer Scar Assessment Scale (POSAS) | at day of discharge (approximately 1 week) and at follow-up visit depending on routine clinical practice (approx. 1-3 months postoperatively)
  Effectiveness parameter: Patient and Observer Scar Assessment Scale (POSAS) The POSAS consists of two parts: a Patient Scale and an Observer Scale. Both scales contain six items that are scored numerically and make up a 'Total Score' of the Patient and Observer Scale. Each item of both scales has a 10-point score, with 10 indicating the worst imaginable scar or sensation. The lowest score is '1', and corresponds to the situation of normal skin (normal pigmentation, no itching etc), and goes up to the worst imaginable. The Total Score of both scales can be simply calculated by summing up the scores of each of the six items. The Total Score will therefore range from 6 to 60. Besides the six items the 'Overall Opinion' of the scar quality is scored separately of both patients and observers. [http://www.posas.org]
Cosmetic outcome | at day of discharge (approximately 1 week) and at follow-up visit depending on routine clinical practice (approx. 1-3 months postoperatively)
  Effectiveness parameter: Evaluation of the wound using VAS (1 worse - 10 excellent)
Pain | at day of discharge (approximately 1 week) and at follow-up visit depending on routine clinical practice (approx. 1-3 months postoperatively)
  Effectiveness parameter: using the visual analogue scale (VAS 1 - 10) at discharge, and at follow-up visit depending on the routine clinical practice.
Satisfaction of the patient | at day of discharge (approximately 1 week) and at follow-up visit depending on routine clinical practice (approx. 1-3 months postoperatively)
  until day of discharge, and at follow-up visit depending on routine clinical practice using VAS (1 - 10).
Handling of the suture material | intra-operatively
  Performance Parameter: questionnaire including different dimensions (knot security, tensile strength, knot run down, tissue drag, stiffness, etc) with 5 evaluations levels (excellent, very good, good, satisfied, poor).

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Leopoldina-Krankenhaus GmbH, Schweinfurt, Bavaria
  - Benedictus Krankenhaus Tutzing GmbH & Co., Tutzing, Bavaria
  - Klinikum der Johann-Wolfgang-Goethe Universität, Department for Pediatric Surgery and Pediatric Urology, Frankfurt am Main, Hesse

REFERENCES:
- [Result] Baumann P, Gumpinger F. Prospective, Observational Study to Assess a New Quick Absorbable Monofilament Suture for Skin Closure in Adults. Journal of Surgery 2021; 9(2):63.
- [Result] Baumann P, Weigel M. Episiotomy Closure After Vaginal Delivery-A Prospective, Single Centre Study Assessing a Novel Fast-Absorbable, Monofilament Suture in Daily Practice. Journal of Surgery 2021; 9(3):121.